CLINICAL TRIAL: NCT05073042
Title: Targeting Diurnal Exercise Timing to Increase Exercise Levels Among Adults With Obesity: A Randomized, Crossover Pilot
Brief Title: Evaluating the Feasibility and Acceptability of Prescribed Diurnal Exercise Timing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20-01292
Record Dates: First submitted 2021-09-08; First posted 2021-10-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: physical activity; exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Morning exercise (Experimental): Participants will have a daily exercise goal, receive nightly surveys, receive weekly emails, and wear a physical activity sensor daily.
  Interventions: Behavioral: Morning exercise goal
- Evening exercise (Experimental): Participants will have a daily exercise goal, receive nightly surveys, receive weekly emails, and wear a physical activity sensor daily.
  Interventions: Behavioral: Evening exercise goal
- Time of choice exercise (Active Comparator): Participants will have a daily exercise goal, receive nightly surveys, receive weekly emails, and wear a physical activity sensor daily.
  Interventions: Behavioral: Time of choice exercise goal
- No exercise period (No Intervention): During the two-week "washout" (i.e., break) periods between the exercise interventions, participants will not have an exercise goal. Participants will continue to receive weekly emails and wear a physical activity sensor daily.

INTERVENTIONS:
Behavioral: Morning exercise goal — Participants will be instructed to walk at a moderate intensity for at least 15 continuous minutes between 5 AM and 10 AM each day.
  Arms: Morning exercise
Behavioral: Evening exercise goal — Participants will be instructed to walk at a moderate intensity for at least 15 continuous minutes between 5 PM and 10 PM each day.
  Arms: Evening exercise
Behavioral: Time of choice exercise goal — Participants will be instructed to walk at a moderate intensity for at least 15 continuous minutes at a time of their choice each day. This time can change day-to-day.
  Arms: Time of choice exercise

SUMMARY:
This pilot study seeks to learn more about people's experiences with being asked to exercise consistently at a specific time of the day (e.g., in the morning) and whether a certain exercise time is most helpful for becoming more active. All participants will be asked to walk for at least 15 minutes per day at a specified time of day (morning, evening, or time of choice) for 3 weeks each (9 weeks of walking total). Each 3-week exercise period will be separated by 2 weeks with no exercise goal. Participants will be emailed a brief survey about barriers/facilitators to exercise each night during the exercise periods and will receive a weekly email that provides support and encouragement for increasing physical activity. Participants will also wear a physical activity monitor on their waist each day during the study to measure physical activity. Participants will complete questionnaires about their experiences at the end of the study.

DETAILED DESCRIPTION:
Performing at least 150 minutes of moderate intensity physical activity per week is associated with many health improvements. Some research suggests that people who exercise at the same time day-to-day perform more physical activity than those who exercise at variable times day-to-day, but it is not yet known if asking people to exercise at the same time day-to-day is helpful for becoming more active and whether there is a specific time of day (e.g., morning vs. evening) that is most helpful. Importantly, it is also not yet known whether people are able and willing to exercise at a specific time day-to-day. This study thus seeks to learn more about how feasible, acceptable, and helpful it is to exercise at an assigned time.

The study will last for 4 months total. Interested participants will be asked to attend an orientation visit at the research center to learn more about the study and will wear a physical activity monitor for 1 week to verify eligibility. Participants who enroll in the study will then complete a 45-minute session with study staff (in person or via videoconferencing) to learn strategies for safely increasing physical and will be asked to walk at a moderate intensity for at least 15 consecutive minutes every day during three, 3-week periods (9 weeks total). Each participant will be asked to perform this walking in the morning (5:00-10:00 AM) for one of the 3-week periods, in the evening (5:00-10:00 PM) for one of the 3-week periods, and at a time of their choice for one of the 3-week periods. Between each 3-week period with a daily exercise goal, there will be a 2-week break period with no exercise goal. Participants will be asked to wear a physical activity sensor on an elastic band around their waist during all waking hours for the full study duration to monitor their physical activity levels. They will also be emailed a survey about their physical activity each night during each of the 3-week exercise periods. Participants will receive a weekly email each week to provide support and encouragement for increasing their physical activity, and to report on how many days they wore the physical activity sensor. Lastly, participants will complete a visit at the research center at the end of the study to complete questionnaires about their experiences.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 65 years of age
* BMI between 30.0 and 50.0 kg/m2
* Able to read and write English
* Home access to the internet via computer or smart phone
* Ability to walk 10 consecutive min without assistance
* Currently performing <50 min/week of moderate intensity physical activity per week (verified via an accelerometer)

Exclusion Criteria:

* Current participation in another formal weight management or physical activity intervention
* Pregnant, <6 month postpartum, or planning to become pregnant in the next 3 months
* Presence of an uncontrolled mental health condition
* Extended absence (e.g., extended vacation) from the Providence area during the study
* Presence of a medical condition for which increased exercise may be contraindicated

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Consent rates | Pre-intervention
  Percent of eligible individuals electing to enroll in the study
Study completion rates | At study completion, an average of 14 weeks
  Percent of consented individuals completing the post-intervention assessment
Physical activity timing adherence rates | Through study completion, an average of 14 weeks
  Percent of moderate intensity physical activity bouts per 3-week condition completed during the assigned time (i.e., 5-10 AM for the morning condition, 5-10 PM for the evening condition)
Acceptability questionnaire | At study completion, an average of 14 weeks
  17-item questionnaire assessing satisfaction with and perceived helpfulness of prescribed physical activity timing overall and specifically in the morning and evening

SECONDARY OUTCOMES:
Average daily physical activity minutes | Through study completion, an average of 14 weeks
  Average daily minutes of moderate-to-vigorous physical activity per week per each 3-week timing condition as measured by a hip-worn accelerometer
Average days per week with at least 15 min of physical activity | Through study completion, an average of 14 weeks
  Average number of days per week with at least 15 minutes of moderate-to-vigorous physical activity per each 3-week timing condition as measured by a hip-worn accelerometer
Barriers and facilitators of physical activity questionnaire | Through study completion, an average of 14 weeks
  Questionnaire administered nightly during each 3-week exercise period that assesses the presence and intensity of several barriers to (e.g., fatigue, scheduling conflicts) and facilitators of (e.g., habit, enjoyment) physical activity.
Preferred physical activity timing questionnaire | At study completion, an average of 14 weeks
  Two self-report questions assessing preferred physical activity timing

CONTACTS AND LOCATIONS:
Overall Officials: Leah Schumacher, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided